CLINICAL TRIAL: NCT03921060
Title: Markers of Osteoporosis in Cystic Fibrosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raksha Jain, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STU 052018-007
Record Dates: First submitted 2019-03-26; First posted 2019-04-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main Study (No Intervention): Up to 100 subjects, both non-CF volunteers and Cystic Fibrosis (CF) patients, will participate in a single study visit that will include a DEXA scan (if not completed as standard of care within 6 months prior to research visit), micro CT, and blood collection.
- Denosomab Sub-study (Experimental): Approximately 10 subjects with CF that have completed the main study and have results which indicate bone disease are eligible to participate in the sub study. Subjects who consent will receive treatment with denosumab (60 mg/ml via subcutaneous injection in the upper arm, upper thigh, or abdomen every 6 months) for up to 5 years. These subjects will be asked to return every 6 months for injections and annually (+/- 6 months) for up to 5 years for a DEXA scan, micro CT, and blood collection.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — treatment with denosumab every 6 months for up to 5 years
  Arms: Denosomab Sub-study

SUMMARY:
Main Study Up to 100 subjects, both non-CF volunteers and Cystic Fibrosis (CF) patients, will participate in a single study visit that will include a DEXA scan, micro CT, and blood collection.

Denosumab (Prolia) Sub study Approximately 10 adult subjects with CF who participated in the main study and have results indicating bone disease will receive treatment with Denosumab for up to 5 years. They will be asked to return annually for repeat DEXA scans, micro CT, and blood collection.

ELIGIBILITY:
Cystic Fibrosis Main Study Inclusion Criteria:

* Must have CF diagnosis confirmed by sweat test or genotype analysis
* Subjects (and parents/legal guardians as applicable) must have the ability to read and write in English

Sub-study Exclusion Criteria:

* No CF diagnosis
* Men or women without osteoporosis
* Less than 18 years of age
* Unwilling to return annually for study visits for up to 5 years
* Unwilling and/or medically unable to take denosumab

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
DEXA results | Looking at single timepoints and well as changes for up to 5 years for those in the sub-study
  Z and/or T scores
Micro CT results | Looking at single timepoints and well as changes for up to 5 years for those in the sub-study
  Trabecular bone volume to tissue volume (BV/TV), cortical and trabecular thickness (Tb.Th, microns), trabecular spacing (Tb.Sp; microns), and structure model index (SMI; index of trabecular rod vs plate-like shape/ stoutness) will be assessed. Change in BV/TV and cortical thickness will be taken to indicate increased/decreased bone mass accrual by microCT.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No